CLINICAL TRIAL: NCT04590833
Title: Feasibility Testing a Randomized Controlled Trial of an Exercise Program to Improve Cognition for T2DM Patients
Brief Title: Feasibility Testing an Exercise Program to Improve Cognition for T2DM Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arkansas, Fayetteville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2005265810
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: cognitive dysfunction; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Experimental)
  Interventions: Behavioral: Supervised walking on a treadmill
- Attention control group (Placebo Comparator)
  Interventions: Behavioral: Supervised stretching exercise

INTERVENTIONS:
Behavioral: Supervised walking on a treadmill — Each participant will be provided with an individualized target heart rate zone based on his/her age. Heart rate during exercise will be measured using a finger pulse oximeter. Following baseline measures, participants will receive instructions on how to use a finger pulse oximeter by a student. For participants who are not physically fit or are just engaging in regular exercise, they will be advised to start walking on a treadmill at a comfortable pace for 5 to 10 minutes at one time.46 Exercise duration and intensity will be progressed from week 3 to week 5, until participants will walk at 40-59% of heart rate reserve based on their age, which will be maintained throughout the study.
  Arms: Aerobic exercise group
Behavioral: Supervised stretching exercise — Following baseline measures, a student will demonstrate the use of a pulse oximeter and stretching movements to these participants. Starting on week 3, participants will do the prescribed stretching exercise 3 times a week, maintaining heart rate below 40% of heart rate reserve during exercise. Stretching will target all major muscle-tendon groups including shoulder, chest, neck, truck, lower back, hips, and legs. It will also involve a slow and constant motion that accounts for any physical limitations and physician-specified precautions
  Arms: Attention control group

SUMMARY:
This proposed study will advance science by providing evidence on the feasibility of a standardized, rigorously designed and delivered exercise program to improve cognition and plasma brain-derived neurotrophic factor (BDNF) levels for individuals with type 2 diabetes. We will also explore how certain genetic variant may influence exercise-induced cognitive improvements and plasma BDNF levels. Findings of the proposed study will establish a comprehensive knowledge base for future research and development of a personalized exercise program for high-risk individuals who are vulnerable to cognitive dysfunction based on their genomic profiles.

DETAILED DESCRIPTION:
The study will pilot-test a 3-month supervised exercise program to improve plasma brain-derived neurotrophic factor (BDNF) levels and domains of cognition that are mostly affected in type 2 diabetes mellitus (T2DM), including memory, processing speed, and executive function, overall and according to genotypes of the BDNF Val66Met variant. T2DM impairs the brain, leading to cognitive dysfunction, which carries substantial lifetime consequences. This highlights an urgent need to find effective therapeutic strategies to improve cognitive function among those with T2DM. Aerobic exercise enhances cognitive function among healthy subjects through increased release of BDNF. BDNF supports survival of existing neurons and promotes growth of new neurons and synapses. Emerging evidence suggests that reduced BDNF levels may exacerbate cognitive dysfunction associated with T2DM. Compared to drug delivery of BDNF, aerobic exercise is a low- cost, safe, and easily accessible path to increasing endogenous BDNF levels. In persons with T2DM, integrity of the blood-brain barrier (BBB) is impaired. Although a growing body of evidence supports the protective role of regular exercise in BBB integrity, very little is known about how resting peripheral BDNF levels may change in response to regular aerobic exercise training after adjusting for BBB permeability among individuals with T2DM. One critical genetic variant that affects cognition in human is the BDNF Val66Met variant. The Met allele interferes with the activity-dependent secretion of mature BDNF among Met carriers. Despite the strong evidence suggesting aerobic exercise has a beneficial effect on cognitive function, significant variability in individual response to exercise training in cognitive outcomes has been reported among Val/Val vs. Met carriers. However, the evidence on how the BDNF Val66Met variant influences cognitive outcomes following an aerobic exercise intervention among individuals with T2DM is currently lacking. A total of 84 participants with T2DM will be randomized 2:1 to receive aerobic exercise intervention (n=56) or attention control (n=28) for 3 months. The study will evaluate the feasibility of the intervention. The study will also evaluate preliminary effectiveness of the supervised exercise program on cognitive function and plasma BDNF levels after controlling BBB permeability. An exploratory aim is to explore the influence of the BDNF Val66Met polymorphism on cognitive outcomes and plasma BDNF levels in response to aerobic exercise intervention. The purpose of this study is well aligned with the National Institute of Nursing Research (NINR) mission to develop personalized interventions that address mechanisms underlying symptoms of illness through symptom science research. Based on the findings of this proposed study, our long-term goal is to develop a personalized exercise program for high-risk individuals susceptible to cognitive dysfunction based on their genomic profiles.

ELIGIBILITY:
Inclusion Criteria:

* Participants eligible for this study will be sedentary adults with no major chronic physical or mental disorders but classified as having low physical activity levels determined by the International Physical Activity Questionnaire.
* Participants must have a documented medical diagnosis of T2DM and must be receiving diabetes care at the time of enrollment.
* Participants must be English-speaking and are able to give informed consent.

Exclusion Criteria:

* include uncontrolled hypertension with resting blood pressure of 160/90 mmHg or higher, having symptoms of coronary ischemia such as chest pain and severe shortness of breath during activities of daily living, loss of consciousness/fainting for any reason, or having any other medical or physical conditions (such as osteoporosis, asthma, spinal cord injury) or symptoms (e.g., pain or swelling in any part of the body) that may interfere with exercise participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-09-24 (Estimated); Study Completion 2023-09-24 (Estimated)

PRIMARY OUTCOMES:
Episodic memory | Three months
  Picture Sequence Memory Test. Test-retest reliability of the test is 0.77. Convergent validity and discriminant validity is 0.69 and -0.08, respectively.
Executive function | Three months
  Dimensional Change Card Sort Test. Test-retest reliability of the test is 0.88. Convergent validity and discriminant validity is -0.51 and 0.14, respectively.
Working memory | Three months
  List Sorting Working Memory Test. Test-retest reliability of the test is 0.77. Convergent validity and discriminant validity are 0.58 and 0.30, respectively.
Processing speed | Three months
  Pattern Comparison Processing Speed Test. The test takes about 3 minutes to compete. Test-retest reliability of the test is 0.72. Convergent validity and discriminant validity is 0.49 and 0.12, respectively.

SECONDARY OUTCOMES:
Plasma BDNF in ng/mL | Three months
  BDNF in plasma will be measured using an ELISA kit.
Fasting blood glucose in mg/dL | Three months
  Fasting blood glucose will be measured using YSI.
HbA1c in percentage | Three months
  HbA1c will be measured using an ELISA kit.
Weight in kilograms | Three months
  Weight will be measured with a health scale.
Height in meters | Three months
  Height will be measured using a stadiometer.
BMI | Three months
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No